

# "Developmentofaneuronalmicroscopeforcellcharacteri zationandmanipulation"

# (NeuronalmicRoscopyforcellbehaviorVioural Examinationandmanipulation)

Acronym: REVEAL

Protocolversionnumber:see1.0Date:09December2020

**Promoter:**IRCCSCa'GrandaFoundationMaggiorePoliclinicoHospital,ViaSforza 28,20122Milan,Italy

Coordinatingcenter: UOC Transfusion Center IRCCSCa'GrandaFoundationOspedaleMaggiorePoliclinico, ViaSforza35, 20122Mil an, Italy

lau Volet.

**PrincipalInvestigator**:Prof.Luca VittorioValenti

# **STATEMENTOFCONFIDENTIALITY**

AllinformationpresentedinthisdocumentwillbeconsideredconfidentialandwillremaintheexclusivepropertyofFondazioneIRC CSCa'GrandaOspedaleMaggiorePoliclinico.Theuseofsuchconfidentialinformationmustbelimitedto the recipient for the agreed purpose and must not be disclosed, published or otherwise communicated tounauthorizedpersons,foranyreason,inanyformwithoutthepriorwrittenconsentofFondazioneIRCCSCa'GrandaOspedaleM ajorPolyclinic.









# **FLOWCHART**

| | Screening | Intervention |
|---------------------------------|-----------|--------------|
| Period | (-t1) | (t1) |
| Enlistment | | |
| informedconsent | - | |
| inclusion/exclusioncriteria | - | |
| Administrationoftheintervention | | |
| Biologicalsamplecollection | | - |

# **LISTOFABBREVIATIONS**

ALS:Automated Lab Solutions GmbH

**THEREIS:**EthicsCommittee

**CEA**:Commissariatàl'énergieatomiqueetauxénergiesalternatives

CI:InformedConsent

**CRF**:CaseReportForm,datacollectionform**EC**:

EuropeanCommunity

ENS: Ecole Normale Supérieure de Lyon GCP: Good Clinical Practic

e, good clinical practice HCC:HepatocellularCarcinoma,

hepatocellularcarcinomaLMU:LudwigMaximilian University

of Munich WUT:PolitechnikaWarszawska





# **TITLEPAGE**

# FLOWCHART LISTOFABBREVIATIONSINDEX1.INTRO DUCTION

1.1 Backgroundandrationale

#### 2. OBJECTIVEOFTHETESTING

- 2.1 Primaryobjective
- 2.2 Secondaryobjective(s).

#### 3. STUDYDESIGN

- 3.1 Studydesign
- 3.2 Inclusioncriteria
- 3.3 Exclusioncriteria

# 4. PROCEDURES RELATINGTOTHESTUDY

- 4.1 Intervention
- 4.2 Randomization
- 4.3 Blindness

# 5. ENDPOINTS

- 5.1 Primaryendpoint
- 5.2 Secondaryendpoint

# 6. DURATION/TIMELINEOFTHESTUDY

- 7. STATISTICALANALYSIS
  - 7.1 Samplesizeanddataanalysis
- 8. ADVERSEEVENTS
- 9. RISK/BENEFITASSESSMENT





e formazione universitaria



#### 10. PRACTICEMANAGEMENT

- 10.1 Datacollectionandmanagement
- 10.2 Regulatoryaspectsandethicalconsiderations
  - 10.2.1 Approvalofthecompetentauthority
  - 10.2.2 ApprovaloftheEthicsCommittee
  - 10.2.3 Informedconsent
- 10.3 Dutiesoftheinvestigator
- 10.4 Studymonitoring
- 10.5 Qualityassuranceofthestudy
- 10.6 Closureofthestudy
- 10.7 Archivingofdocuments
- 10.8 Disclosureofinformationregardingscientificdiscovery
  - 10.8.1 Confidentiality
  - 10.8.2 Publications
- 10.9 Intellectual property rights on the study results
- 11. Indemnityandcompensationincaseofdamages
- 12. FinancialArrangements
- 13. ConflictsofInterestDisclosure
- 14. References

#### 1. INTRODUCTION

#### 1.1 Backgroundandrationale

Hepatocellularcarcinoma(HCC)isthemostcommontypeofprimarylivercancerandisaleadingcause of cancer-related death worldwide. The prognosis of HCC remains poor, with yearsurvivalrateof18%(1).RiskfactorsforHCCincludeviralinfection,autoimmunehepatitis,chronicalcoh metabolic fatty ol use liver disease. obesity. and diabetes mellitus Furthermore, alterations and chronic inflammation of the microenvironment can facilitate the transformation of the microenvironment can facilitate the microenviro onofnormalliverstemcellsintoprecanceroustumorstemcells(3). Alltheseunderlyingpathogenicstimulic aninduceaspectrumofgeneticandepigeneticmodifications, which are involved in the cell cycle, cell growth andregulation of adhesion. Therefore, heterogeneity and tumor priming potential arise from a combination nofbothendogenous and exogenous factors (4). In particular, he patocellular carcinomais an extraordinari lyheterogeneous diseased ue to the morphological and histological diversity of livercell types, and such intrinsical diversity of livercell types, and such intrinsical diversity of livercell types. atumoralheterogeneityrepresentsamajorchallengefortumorcharacterizationandtherapeuticmanage mentofpatientswithHCC.

Currentinvitromodels, based on conventional hepatoma and hepatocarcinoma cell lines, fail to recapitulate key characteristics of tumortissue such as three-dimensional tissue architecture, cellular heterogeneity, and cell-cell interactions. Organoids, which are 3D cellular structures generated from both induced pluripotents tem cells and adult tissue-

residentstemcells, have recently been exploited to overcome the limitations of 2D cell culture systems, emerging aspowerful tools for studying human diseases (5, 6). This is possible as they are able

stablypreservethegeneticinformationoftheautologoustissueandmimicthepathologicalstateofthetissu eitself.

These structures will be the basis for developing a new and promisingmethodology of microscopy, called "neuronal", which is strongly based on neural networks capable of perception, interpretation, inference, prediction, decision, and action.

#### 2. OBJECTIVE/HYPOTHESISOFTHEEXPERIMENT

Theaimoftheproject, within which this clinical study is part, is to validate the ability of a "neuronal" microscope to decipher the molecular

mechanismsattheoriginofcancer, especially by addressing the problem of biological heterogeneity. Molecular characterization of tumor cell subtypes at the single-cell level has the potential to resolve the temporal order of events governing the developmental trajectories of livercancer. Thanks to the neuronal microscopeable

to select individual cells, we intend to identify and isolate cells at different points of the trajectories that lead from the content of t



Polo di ricerca, cura e formazione universitaria









#### omthenormalstatetothe









e formazione universitaria

tumor("past,presentandfuture").

Morespecifically, the scientific projectaims to develop a "cell-

harvestingneuronalmicroscope"thatwillallowincombinationwithbiological analyses (proteomics, genet ics, etc.) to characterize the cellular heterogeneity known to cause liver cancer. The challenge is to develop this new molecular imaging technique which can potentially reveal new cellular mechanisms at the origin of a disease.

Todemonstratethat, this neuronal microscopy can lead to understanding the cellular origin of a disease, it will be used to decipher, identify and predict the state of cells originating from liver tumors derived from patients and mouse models of this disease.

# 2.1 Primaryobjective

TheprimaryobjectiveofthestudyconductedattheFondazione IRCCS Ca' Granda Ospedale Maggiore Policlinicoistogenerateandcharacterizethree-dimensionalcell culture models,calledorganoids,ofthemainlivercellpopulations,inordertoimitatetheearlystages of human carcinogenesisand then analyze the onsetof HCC, to identifythe specific mechanismsinvolvedinhepatocellularcarcinoma.

# 2.2 Secondaryobjectives

- 1. Liverorganoids(normal,pre-tumorortumor) are used to "train" theneuronal microscope in order to distinguish various cells ubtypes within heterogeneous cultures and recognize pre-neoplastic cells able to initiate the transition from a normal state to a tumor state.
- 2. On thisbasis, a "singlecell sampling" system will be developed that will allow us to detect and collect different subtypes of liver cells that are expected to be come can cerous and to analyze them before the tumor manifest sitself.

#### 3. STUDYDESIGN

#### 3.1 Studydesign

Interventional, with the collection of biological, non-pharmacological, monocentric material.





# **RESPONSIBILITY**(roleofthepromoterandcollaborators)

| Operationalunit | Participantname | Roleandfunctionsinthefirm |
|---|---|---|
| Department of TransfusionMedicineandHematolo gy, Fondazione IRCCSCa' Granda Ospedale MaggiorePoliclinico | Dr.DanielePrati Prof.LucaValenti(principalinvestigator) | Samplerecruitmentandcharacterization;<br>Isolation and generation<br>oforganoids,spheroidsandtissues;Ch<br>aracterizationoforganoidsbygeneand<br>proteinexpression |
| | | Dataanalysis |

# Internalcollaborations:

| Operationalunit | Participantname | Roleandfunctionsinthefirm |
|---|---|---|
| UOCGeneralSurgeryandLi<br>verTransplants,<br>Fondazione IRCCS Ca' Granda<br>OspedaleMaggiorePoliclinico | Prof.GiorgioRossi | Reportingofeligiblepatientsandsampl echaracterization |
| UOCScientificDirectionFondazio<br>ne IRCCSCa' Granda<br>OspedaleMaggiorePoliclinico | Dr.StefanoGatti | Reporting of eligible patients, sample characterization and supportincell isolation protocols |

#### Externalcollaborations:

| Collaboratingbody | Roleandfunctionsintheproject |
|---|---|
| Commissariatàl'énergieatomiqueetauxénergiesalternatives,France(CEA) | Development of the 2D neuronal scanning lens-free microscopeandprototypingofthe3Dneuronalmicroscope;valida tionofthemicroscopeprototypesthroughtheuseofhumanandmu rinesamplesgeneratedrespectivelyattheFoundationandENSLy on |
| Iprasense,France | Technicaldevelopmentandimplementationofthelens-free neuronalmicroscope |
| EcoleNormaleSupérieuredeLyon,France(ENS) | Generation of mouse models of liver disease; processing and is olation of samples generated at the Foundation; sequencing and transcriptomic analysis of single cells to generate cell trajectories |

ISTITUTO DI RICOVERO E CURA A CARATTERE SCIENTIFICO DI NATURA PUBBLICA Via Francesco Sforza, 28 - 20122 Milano Tel. 02 5503.1 - www.policlinico.mi.it - CF e P.I. 04724150968





e formazione universitaria

| LudwigMaximilianUniversityofMunich,Germany(LMU) | Proteomicandmulti-omicanalyzesofcellandorganoidclusters |
|---|---|
| AutomatedLabSolutionsGmbH,Germany(ALS) | Developmentandvalidationofthelens – freeneuronalmicroscope; creationoftheprototypefortheis olationofsinglecells |
| PolitechnikaWarszawska,Poland(WUT) | Metrological evaluation and validation of the developed 2Dand 3D microscopes, through the design and production ofcalibrationsamplesusing3Dprintingtechnology |

# 3.2 Inclusioncriteria

Adultpatientsundergoingsurgicalcholecystectomy, liverresection for hepatocellular carcinoma or whole liver explants, who have given consent to participate in the study, will be included.

#### 3.3 Exclusioncriteria

Patientswhoarepositiveforchronicviralhepatitis(HCV-RNAandHBsAg)willbeexcluded.

#### 4. PROCEDURESRELATINGTOTHESTUDY

#### 4.1Intervention

IncollaborationwiththeLiverTransplantUnit of Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, wastetissues amples will be collected from patients undergoing chole cystectomy, liverresection for hepatocellular carcinoma (both intra-tumoral and extra-

tumoraltissues)ortakenfromexplantedwholelivers.

This will allow us to isolate cells and generate organoids starting from the three conditions of interest to us:

- 1) normallivertissues(cholecystectomy);
- 2) diseasedliver(extra-tumoralparenchymaandliverexplants);
- 3) hepatocellularcarcinoma.

Weaimtocollectupto 1 Oindependents amples pertissue type.

To validate the heterogeneity obtained in vitro using organoids, mono- and multi-lineage liverspheroidswillbegeneratedbyexploitingpreviouslyestablishedhepatomacelllines(11),namely:phenoty pically differenthepatomacelllines (HepG2andSNU398cells)





andprimarycelllinesrepresentativeoftumorheterogeneity(HCC-1,HCC-2,HCC-3,generatedwithin thestudy"ImpactoftheI148MvariantofthePNPLA3geneontheregulationofretinolmetabolismand activation of human hepatic stellate cells", Opinion No. 29\_2016 and 29\_2016bis, proceedings300/2016),culturedin96-wellplates.

Tostudytheroleofspecificgeneticpathwaysinregulatingtumorheterogeneity, wewillknockdowngenesof interestforHepG2hepatomacells. Toregulatetheexpressionofspecificproteinsincellular models, wewillu sespecificantisenseoligonucleotides (morpholinos: MPO, GeneTools) that block protein translation, or MPO that does not recognize any mRNA sequence as a control.

The biopsy fragments or fragments obtained from surgical resections will be transported in Celsior perfusion solution at 4°C and will be processed at the Translational Medicinel aboratory in the shortest possible time to isolate liveror ganoids. The tissues will be mechanically fragmented into small pieces, avoiding reducing them to single cells; this will increase the formation efficiency of the organoids. Then the fragments will be further subjected to enzymatic digestion with a solution containing Collagenase and DN as eat 37°C. The cell clusters obtained from enzymatic digestion will be included in reduced growth factor Matrigel. Once the Matrigel has polymerized, the complete culture medium to

growliverorganoidswillbeadded.Isolationsobtainedfromnormaltissueswillbeculturedinmediumcontaining:AdvancedDMEM/F12supplementedwith1%N2and1%B27(bothfromGIBCO),1.25mMN-Acetylcysteine(Sigma),10nMLeu-

Gastrin(Sigma),50ng/mlEGF(Peprotech),1 $\mu$ g/mlRSPO1(Peprotech),100ng/mlFGF10(Peprotech),25 ng/ml HGF (Peprotech), 10 mM Nicotinamide (Sigma), 5  $\mu$ M A83.01 (Peprotech), and 10  $\mu$ M Forskolin(Peprotech).Inordertoincreasetheisolationefficiencyoftheorganoidsforthefirstfewdays,25ng/ml Noggin (Peprotech), 100 ng/ml Wnt3a (peprotech) and 10  $\mu$ M Rock inhibitor Y27632 (Peprotech) willbeaddedtothemedium.Isolationsobtainedfromtumortissueswillbedivided and culturedinclassicalmediumor

intumoroidmediumcontaining:AdvancedDMEM/F12supplementedwith1%N2and1%B27(both from GIBCO), 1.25 mM N-Acetylcysteine(Sigma), 10 nM Leu-Gastrin (Sigma), 50 ng/ml EGF(Peprotech),100ng/mlFGF10(Peprotech),25ng/mlHGF(Peprotech),10mMNicotinamide (Sigma), 5  $\mu$ M A83.01(Peprotech), 10  $\mu$ M Forskolin (Peprotech),and 3 nM dexamethasone(Sigma)(8).

The samples isolated at the Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico will be sent to the ENS in Lyon, that incollaborationwithCEA will develop the transcriptomicanalysis on both whole humanorganoids and isolated cells, using the neuronal microscope.

CEA, through the use of human and murine cells amples is olated at the Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico and ENSLyon respectively, will develop the 2D and 3D imaging platforms. LMU in collaboration with CEA will develop proteomicanalysis both on whole human organoids and on is olated cells using the neuronal microscope.

ISTITUTO DI RICOVERO E CURA A CARATTERE SCIENTIFICO DI NATURA PUBBLICA Via Francesco Sforza, 28 - 20122 Milano Tel. 02 5503.1 - www.policlinico.mi.it - CF e P.I. 04724150968





e formazione universitaria

#### 5. ENDPOINTS

# 5.1 Primary Endpoint

Isolation of epithelial cells in order to generate models of major hepatocellular carcinoma cellpopulations in a three-dimensional culture, called liver organoids, and their molecular characterization of the generated models.

# 5.2SecondaryEndpoints

- $\cdot$  Knowledgeofthebehavioralandmorphological differences between physiological and tumor hepatocytes;
- · Knowledgeofthemolecularmechanismsunderlyingcellularlevelobservationsexploiting "o mics" technologies and CRISPR-Cas9genetic engineering.

#### 6. DURATION / TIMELINE OF THE STUDY

Month and year of study start: 01/2021

Monthand year of enrollment closure: 01/2024

Month and year of studyend: 01/2025

The study will have a duration of 48 months. In the first three years we expect to enroll approximately 30 subjects inaccordancewiththeinclusioncriteria.

# **PROJECTGANTT**

| Intervention | Period(months) | | | |
|------------------------------|----------------|-------|-------|-------|
| | 1-12 | 13-24 | 25-36 | 37-48 |
| Enlistment | - | - | | |
| Informedconsent | - | - | - | |
| Inclusion/exclusion criteria | - | - | - | |
| Generationoforganoids | - | - | - | |











| Evaluationofgeneexpressioninliveror | <br> |
|-------------------------------------|------|
| ganoids | |







e formazione universitaria

| Evaluationofspecificliver proteinsinliverorganoids | <br> | | |
|----------------------------------------------------|------|---|---|
| Datacorrelationanalysis | - | - | - |

#### 7. STATISTICANALYSIS

# 7.1 Samplesizeanddataanalysis

Previously published works (7,8,9,10) have highlighted that the generation efficiency of liver and the state of the stat

organoidsis approximately 90% starting from surgical resections and 33% from biopsies (7,8). Considering these estimates, in order to isolate at least 6 independent organoid cultures of each type of condition of interestinour study, it is estimated to recruitatle ast 30 donors (10 for each condition studied). The intentisto obtain replicates for an alyses with a sufficient representation of the different stages of liver damage (normal liver, inflammation / fibrosis and hepatocarcinoma) and to be able to map the eimpact of the most common hereditary genetic variants (present in at least 20% of individuals) in the population.

The main analyses will be conducted from cell cultures is olated from a single individual. Given the descriptive nature of mapping cellular phenotypes and gene expression, and the large number of organoids (>  $10^3$ ) and cells (>  $10^9$ ) from a single individual, we will have sufficient statistical power (> 80%) to identify and analyzes pecific cellular subsets representing > 1% of the population over all.

# 8. ADVERSEEVENTS

The project does not involve the administration of drugs or other substances or adhoc invasive intervention soutside of normal clinical practices. Therefore, no adverse events are expected.

# 9. RISK/BENEFITASSESSMENT

The study does not predict an immediate benefit for the donors, but the results of this trial will have the potential to lead to a decoding of the mechanisms at the origin of tumor development, resolve the temporal order of the events that regulate the evolutionary trajectory, under stand the progression, characterization and improve the therapeutic management of patients.





# 10. PRACTICEMANAGEMENT

# 10.1 Datacollectionandmanagement

For each participant will be assigned a unique code upon enrollment. The file associating theparticipant'scodewiththerelevantidentificationdatawillbestoredseparatelyonacomputer protected with a password. The study database will be protected with a different password and accessible only to staff designated by the principal investigator. The unique code will be used to prevent that unauthorized individual will be able to discover the identity of the enrolled patient. Only designed investigators will be able to know the identity of the enrolled subjects.

Regardingdatastorage:datathat can be made publicly accessible,to all partnerswillberequiredtouseanopenaccessrepository,linkedtothetoolsproposedbytheEuropeanCommun ity(e.g.OpenAIRE)toensureaccesstopublicationsandabibliographicmetadataarchiveinastandardformat,i ncludingtheinformationrequiredbytheEC.

# 10.2 Regulatoryaspectsandethicalconsiderations

#### 10.2.1 ApprovaloftheCompetentAuthority

Inaccordancewithcurrentregulations, the principal investigator must obtain approval from the appropriate Competent Authority before starting the clinical study.

This study will be conducted in accordance with the rules of the ICH/GCP (International Conference of Harmoniz ation/Good Clinical Practice) and all applicable laws, including the Declaration of Helsinki of June 1964, as a men ded by the latest World Medical Association General Assembly in Seoul, 2008.

# 10.2.2 Approvalof the Ethics Committee

Theinvestigatormustensurethattheprotocolhasbeenseenandapprovedbythelocalindependent Ethics Committee (EC) beforestartingthestudy.

#### TheEC

must also review and approve the informed consent (IC) formand all written information received from the patient prior to enroll mention the study.

If it is necessary to modify the protocol and/or the IC during the study, the investigator will be the guarant or and therefore the person in charge of ensuring the review and approval of this modified document according to the EC's request.

The content of the sechanges will be implemented only after the EC has approved them. Until that time, it will be enecessary to refer to the previous version of the already approved document.







# 10.2.3 InformedConsent(IC)

Theinvestigatororotherstaffdesignedbythe

investigatorshouldinformpeopleaboutallaspectsandproceduresofthestudy.

The process for obtaining informed consent must comply with current regulatory procedures. The investigation of the process of tor(ordesignatedcollaborator)andthesubjectmustdateandsigntheinformedconsentformbeforethat thepatientinitiatesanystudy-related procedures. The subject will receive a copy of the CI dated and signed both parties: the original will be kept by copy archivesdesignatedforstudy. Neither the investigator nordesignated personnels hould in anyway exertany coercion or influence on a subject to participate or continue to participate in the study. Asubject's decision to participate in the study must be completely voluntary. The investigator and designate dpersonnelshouldemphasizetothesubjectthathemaywithdrawconsentatanytimewithoutpenaltyorlos sofanybenefitstowhichhemaybeentitled.

Writtenororalinformationrelatingtothestudy, including the written consent form, must not contain anyling uistic expression that forces the subject to (even apparently) waive his or her legal rights, or that would exoner at ethe investigator, the institution or the sponsor from liability for negligence.

#### 10.3 Dutiesoftheexperimenter

Inaccordancewithapplicablelocalregulations, the investigator must send periodic reports regarding the progress of the study in his center to the EC and notify the EC of the closure of the study. Periodic reporting and closure notification are part of the investigator's responsibilities.

# 10.4 Studymonitoring

In accordance with applicable regulations and good clinical practice (GCP), the clinical monitor must visit or contactthe center periodically. The duration, nature and frequency of such visits/contacts depend on the frequencyof recruitment, the quality of the documents held by the center and their adherence to the protocol.

Throughthesecontacts, the monitor must:

- monitorandevaluatetheprogressofthestudy
- · examinethedatacollected
- $\cdot conduct verification of the source document\\$
- identifyeachproblemanditssolutions







Thepurposes of the monitoring activity are to verify that:

- · the rights and welfare of the subject are respected
- ·The study data are accurate, complete, and can be verified from the original documents
- · the study is conducted in accordance with the protocol and any approved a mendments, GCP and applicable regulations

# Theinvestigatormust:

- · giveto the clinical monitordirectaccesstoallrelevantdocumentation
- $\cdot dedicate part of his and his staff's time to the clinical monitor to discuss the monitoring results and any other possible aspects. \\$

#### Theclinical

monitors hould also contact the center prior to the start of the study to discuss the protocol and data collection procedures with the staff.

# 10.5 Qualityassuranceofthestudy

As Promoter, Fondazione IRCCS Ca'Granda, Ospedale Maggiore Policlinico can carryouta quality controlche ckonthest udyatits discretion. In this case, the investigator must allow the clinical monitor direct access to all relevant documentation and dedicates ome of his or her time and staff to the review er to discuss the monitoring results and any other aspects of the study.

Furthermore, Regulatory Authorities can carry out in spections. In this case, the investigator must grant the inspector direct access to all relevant documentation, and dedicate part of his time and staff to the inspector to discuss the monitoring results and any other aspects of the study.

#### 10.6 Closureofthestudy

At the time of study closure, the monitor and the investigator must activate a series of procedures:

- reviewallstudydocumentation
- · reconcilestudydata
- · reconcileallclarificationreports.





# 10.7 Archivingofdocuments

Inaccordancewithcurrentnationalregulations, the investigator must keep acopy of all documentationands to reitinadry and safeplace after the study is closed.

# 10.8 Disclosureofinformationregardingscientificdiscovery

# 10.8.1 Confidentiality

Theinvestigatorandotherpersonnelinvolvedinthestudymustprocessallinformationrelatingtothestudy(including theprotocol,dataobtainedandalldocumentationproducedduringthestudy)andmustnot use suchinformation, dataor reportsfor purposesother than thosedescribed inthe protocol.

Theserestrictions do not apply to:

- 1) informationthatbecomes publicly available, not due to negligence on the part of the investigator or his staff:
- 2) information requiring confidential disclosure to CE for the sole purpose of evaluating the study;
- 3) informationthatmustbedisclosedinordertoobtainappropriatemedicalcareforastudy subject.

# 10.8.2 Publications

TheIRCCSCa'GrandaFoundation,OspedaleMaggiorePoliclinicoisthesoleownerofthedata.Awebsitededicated totheprojectwillbebuiltwithprivatesectionsthatwillservetheprojectpartnersas update and exchange channels, as well as to build a data archive to be used in the post-projectexploitation phase. The public section will contain the project description (e.g. objectives, partners,fundingsource,etc.),publishedarticlesandongoingwork.Thescientificdirectorofthestudywillwritea final report and make the results public at the end of the study. The data will be made publicanonymouslyandpresentedasrequiredinaggregatemode.InaccordancewiththeprovisionsoftheGrant Agreement,thedisseminationoftheresultswilltakeplaceassoonaspossible,byappropriatemeans,includings cientificpublications.

# 10.9 Intellectual property rights on the study results

Most data will be associated with results that may have commercial or industrial protection potential and therefore cannot be made accessible for verification and re-use generally due to intellectual property protection measures.

However, relevant data necessary for verifying results published in scientific journals can be madeaccessibleonacase-by-casebasis.





 $A Consortium Agreement will be negotiated and signed by all parties in order to specify, among other things, the terms and conditions relating to ownership, access rights, exploitation of the background and results as well as the dissemination of the results, in accordance with the grant agreement and Regulation <math>n^2 1290/2013$  of 11December 2013. The consortium agreement will be based on the DESCAHorizon 2020 Model Consortium Agreement with the necessary adaptations considering the specific context and parties involved in the project and will be based on the following principles:

- · Theparties will identify the knowledge, information, data (of any formornature), know-how, technical material and/or assets protected by industrial and/or intellectual property rights or susceptible to protection, (Background) held and/or developed in any capacity independently by each of the Parties at a time prior to the start of the Project which they will make available for the implementation of the project and will evaluate their availability for access rights with regard to the rights of pot ential third parties on such background to the extent that this information is known to the respective party at the time of the assessment;
- $\cdot \ Ownership of results, including joint results generated by two or more parties, will go to the party or parties that generated such results;$
- · The proprietary parties will take all appropriate measures to protect the results susceptible to commercial or industrial exploitation, in particular through intellectual property rights, where appropriate;
- · The parties will use reasonable efforts to exploit and disseminate the results, directly or indirectly, for example by licensing such results;
- Each party will grant the other parties access rights (through licenses) to its Background and the resultsgenerated during the Project, only if strictly necessary for the implementation of the project itself and/orfortheexploitationoftheresultsofsuchotherparties(onfairandreasonableterms).

#### 11. INDEMNITYANDCOMPENSATIONINCASEOFDAMAGES

In the event of unwanted events or any damage that may arise from participation inresearch, our Institute's Insurance Policy is also extended to cover individual sparticipating in research projects.

# 12. FINANCIALAGREEMENTS

The costs of study procedures exceeding normal clinical practice will be entirely covered by the funds deriving from the Horizon 2020-Europe EU financing.





# 13. DISCLOSURESONCONFLICTSOFINTEREST

Theinvestigators declare no conflicts of interest.

# 14. REFERENCES

- 1- Yarchoan M. et al. 'Recent developments and the rapeutic strategies against he patocellular carcinoma'. Cancer Res. 2019
- 2- YangJDetal.'Hepatocellularcarcinoma:Aglobalview'.NatRevGastroenterolHepatol,2010
- 3- Plaks V. et al. 'The cancers tem cell niche: howes sentialisthen ich ein regulating stemness of tumor cells?'. Cell Stem Cell, 2015
- 4- LawsonDAetal.'Tumorheterogeneityandmetastasisatsingle-cellresolution'.NatCellBiol,2018
- 5- CleversH.'ModelingDevelopmentandDiseasewithOrganoids'.Cell,2016
- 6- FatehullahA.etal.'Organoidsasaninvitromodelofhumandevelopmentanddisease'.NatCellBiol,20
- 7- HuchM,GehartH,vanBoxtelR,HamerK,BlokzijlF,VerstegenMM,EllisE,vanWenumM,Fuchs SA, de LigtJ, vande WeteringM, SasakiN, Boers SJ,Kemperman H,de JongeJ ,ljzermans JN,NieuwenhuisEE,HoekstraR,StromS,VriesRR,vanderLaanLJ,CuppenE,CleversH.Long termcultureofgenome-stablebipotentstemcellsfromadulthumanliver.Cell2015Jan 15;160(1-2):299-312.doi:10.1016/j.cell.2014.11.050.
- 8- Broutier, L., Mastrogiovanni, G., Verstegen, M. et al. Human primary livercancer-derived organoid cultures for disease modeling and drugscreening. Nat Med 23, 1424-1435 (2017). https://doi.org/10.1038/nm.4438
- 9- NuciforoS,Fofanal,MatterMS,BlumerT,CalabreseD,BoldanovaT,PiscuoglioS,WielandS, RingnaldaF,SchwankG,TerraccianoLM,NgCKY,HeimMH.OrganoidModelsofHumanLiverCancersDerivedfr omTumorNeedleBiopsies.CellRep.2018Jul31;24(5):1363-1376.doi:10.1016/j.celrep.2018.07.001.
- 10- Sorrentino, G., Rezakhani, S., Yildiz, E. et al. Mechano-modulatory synthetic niches for liver organoid derivation. *Nat Commun* 11, 3416 (2020).
- 11- PingitoreP,SasidharanK,EkstrandM,PrillS,LindénD,RomeoS.HumanMultilineage3DSpheroidsasaM odelofLiverSteatosisandFibrosis.IntJMolSci.2019;20(7):1629.Published2019Apr2.doi:10.3390/ijms 20071629



Via Francesco Sforza, 28 - 20122 Milano

